CLINICAL TRIAL: NCT07133152
Title: From Codification to Valorisation: a Medico-economic Analysis of Clinical Pharmacy Activities Integrated Into Patient Pathways.
Brief Title: Medico-economic Analysis of Clinical Pharmacy Activities
Acronym: COD-AMAP
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5534
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Stroke Geriatrics Acute Coronary Syndrome Orthogeriatric
Keywords: Clinical Pharmacy; Medico-economic analysis; Iatrogenic; Codification; Valorisation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (8):
- Post-stroke - Active group: Patients hospitalised after a stroke and benefiting from clinical pharmacy activities on their inpatient unit.
  Interventions: Other: Adverse events
- Post-stroke - Comparator group: Patients hospitalised after a stroke and without any clinical pharmacy activities during their hospitalisation.
  Interventions: Other: Adverse events
- Geriatrics - Active group: Patients hospitalised in geriatric settings and benefiting from clinical pharmacy activities on their inpatient unit.
  Interventions: Other: Adverse events
- Geriatrics - Comparator group: Patients hospitalised in geriatric settings and without any clinical pharmacy activities during their hospitalisation.
  Interventions: Other: Adverse events
- Post-Acute Coronary Syndrome - Active group: Patients hospitalised after an Acute Coronary Syndrome and benefiting from clinical pharmacy activities on their inpatient unit.
  Interventions: Other: Adverse events
- Post-Acute Coronary Syndrome - Comparator group: Patients hospitalised after an Acute Coronary Syndrome and without any clinical pharmacy activities during their hospitalisation.
  Interventions: Other: Adverse events
- Orthogeriatric - Active group: Patients hospitalised in an orthogeriatric pathway and benefiting from clinical pharmacy activities on their inpatient unit
  Interventions: Other: Adverse events
- Orthogeriatric - Comparator group: Patients hospitalised in an orthogeriatric pathway and without any clinical pharmacy activities during their hospitalisation.
  Interventions: Other: Adverse events

INTERVENTIONS:
Other: Adverse events — During patient follow-up (hospitalisation + 6 months post-hospitalisation), adverse events will be collected from the patient's computerised medical record (available at the hospital) and by means of a questionnaire carried out by telephone with the patient at 3- and 6-months post-hospitalisation.

SUMMARY:
In recent years, the deployment of clinical pharmacy activities in France has undergone rapid change as a result of the work carried out by the French Society of Clinical Pharmacy (SFPC), organisational innovations (iatrogenic day hospital, city-hospital pathway) and new regulations (adaptation and renewal of prescriptions by hospital pharmacies). This transformation is causing disparities between hospitals in the deployment of clinical pharmacy activities and a lack of clarity in the activities of each.

At the same time, the traceability of these clinical pharmacy activities is a major strategic challenge, as it meets regulatory requirements (pharmaceutical analysis linked to dispensing), safety requirements (pharmaceutical interventions, reconciliation of drug treatments), financial requirements (day hospital, medical and rehabilitation care, outpatient consultations) and quality requirements (reglutory indicators, mandatory certification).

Some healthcare institutions have launched local initiatives to code their clinical pharmacy activities themselves. These experiments have demonstrated the need to standardize coding across French healthcare institutions, in order to bring it into line with current guidelines (French Health Authority - HAS - guidelines, good clinical pharmacy practice, decree) and the coding rules of the common classification of medical acts. The ultimate aim of such coding is to qualify, in the long term, for financial recognition of clinical pharmacy activities via the Health Insurance System. To meet this need, in March 2023 OMEDIT PACA-Corse published a coding guide for clinical pharmacy activities, validated by the SFPC and deployed to date in a number of French establishments.

Based on national coding, the investigators propose to carry out a medico-economic analysis using observational data, in order to assess the efficiency of integrating clinical pharmacy activities into patient care pathways. The aim of this study is also to initiate a process of reflection to define the pharmaceutical costs associated with clinical pharmacy activities. The investigators hypothesize that the costs of implementing clinical pharmacy (hospital pharmacist salary) will be covered by the costs avoided in terms of adverse events.

A single-centre, prospective, non-interventional and comparative cohort study will be carried out in 4 different care pathways with 2 different sites targeted for each pathway: one site carrying out clinical pharmacy activities with patients as part of routine care (active group) and one site carrying out no clinical pharmacy activities with patients as part of routine care (comparator group).

The study takes place in the same way in each of the 4 pathways, with 3 distinct phases:

Phase 1: Collection of routine care data during hospitalisation:

* In the active group: no research-related procedures are carried out on the patient. The patient benefits from the clinical pharmacy activities offered as part of routine care. The pharmacist records the time spent with the patient for each clinical pharmacy activity performed during the hospital stay.
* In the comparator group: no research-related activities are performed on the patient. Patients benefit from the routine care pathway defined in their hospital ward.

Phase 2: Collection of routine care data at 3- and 6-months post-hospitalisation:

- In the active group and in the comparator group: consultation of the computerised patient record to collect adverse events related to drug management that occurred at 3- and 6-months post-hospitalisation (emergency room visits, hospitalisation, drug-related iatrogenicity);

Phase 3: Telephone call to the patient 3- and 6- months after hospitalisation:

- In the active group and in the comparator group: evaluation via a questionnaire of adverse events related to drug management which occurred in the 6 months post-hospitalisation (emergency room visits, hospitalisation, drug-related iatrogenicity, consultation with the treatment physician). The call at 3 months is optional.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Admitted to the hospital during the 2 months of recruitment
* Hospitalized in one of the following care pathways: post-stroke, geriatrics, post-acute coronary syndrome, orthogeriatric.

Exclusion Criteria:

* Patients who have expressed their opposition to the study;
* Patient under curatorship, guardianship or legal protection;
* Patients unable to express their non-opposition;
* Person deprived of liberty by a judicial or administrative decision;
* Person under compulsory psychiatric care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients, medical pathways (post-stroke, geriatrics, post-acute coronary syndrome, orthogeriatric).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cost/efficiency ratio | At 3-monts post-hospitalisation (facultative) At 6-months post-hospitalisation (mandatory)
  Numerator: production costs of clinical pharmacy activities per patient (expressed in Euro, from hospital pharmacist's salary) Denominator: adverse events avoided (expressed in adverse events number, difference in frequency per patient between the comparator group and the active group)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Bron, France
  - Hospices Civils de Lyon - Hôpital Renée Sabran, Hyères, France
  - Hospices Civils de Lyon - Hôpital Edouard Herriot, Lyon, France
  - Hospices Civils de Lyon - Hôpital de la Croix-Rousse, Lyon, France
  - Hospices Civils de Lyon - Hôpital Lyon Sud, Oullins, France
  - Hospices Civils de Lyon - Hôpital des Charpennes, Villeurbanne, France